CLINICAL TRIAL: NCT05785325
Title: RC48-ADC Combined With Bevacizumab in HER2-positive Advanced Colorectal Cancer：a Single-arm, Non-randomized, Single-center Trial
Brief Title: RC48-ADC Combined With Bevacizumab in HER2-positive Advanced Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-010
Record Dates: First submitted 2023-03-13; First posted 2023-03-27 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2022-12

CONDITIONS: Colorectal Cancer
Keywords: RC48-ADC; Her2-positive; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RC48-ADC plus Bevacizumab (Experimental): Administer RC48-ADC intravenously in combination with bevacizumab 5mg/kg once every two weeks. Medication must be discontinued until disease progression, intolerable toxicity, informed consent is withdrawn, or investigator judgment is made.
  Interventions: Drug: RC48-ADC plus Bevacizumab

INTERVENTIONS:
Drug: RC48-ADC plus Bevacizumab — Administer RC48-ADC intravenously in combination with bevacizumab 5mg/kg once every two weeks.

SUMMARY:
A phase II clinical study of RC48-ADC combined with Bevacizumab as late-line treatment in patients with HER2-expressed metastatic colorectal cancer. A total of 30 patients are planned to be enrolled.

DETAILED DESCRIPTION:
This is a single-arm, non-randomized, single-center trial. Enroll 30 patients with HER2-expressed metastatic colorectal cancer and failure of standard therapy. Divide into 2 cohorts, including 10 patients with low HER2 expression (IHC 2+/FISH negative) and 20 patients with high HER2 expression (IHC 2+/FISH positive or IHC3+). Administer RC48-ADC intravenously in combination with bevacizumab 5mg/kg once every two weeks. Medication must be discontinued until disease progression, intolerable toxicity, informed consent is withdrawn, or investigator judgment is made. The primary endpoints is objective response rate (ORR), and secondary endpoints are progression-free survival (PFS), overall survival (OS), and adverse effects (AE).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or above, male or female;
2. Advanced inoperable colorectal cancer confirmed by pathology;
3. At least 1 measurable lesion meeting RECIST v1.1 criteria;
4. Patients who had received at least oxaliplatin, irinotecan, and fluorouracil for advanced or metastatic disease progressed or were intolerant were admitted to the study; Patients who had previously received anti-HER2 therapy such as trastuzumab and lapatinib were allowed to be included;
5. ECOG PS: 0-2 points;
6. Patients with HER2 expression: IHC results 2+ or 3+.
7. Predicted survival ≥12 weeks;
8. Women of childbearing age must already be using reliable contraception or have had a pregnancy test (serum or urine) with negative results within 7 days prior to inclusion and be willing to use an appropriate method of contraception during the trial period and 8 weeks after the last test drug administration. For males, consent is required to use an appropriate method of contraception or surgical sterilization during the trial period and 8 weeks after the last administration of the trial drug;
9. The subjects voluntarily joined the study and signed the informed consent. The subjects had good compliance and cooperated with follow-up visits.

Exclusion Criteria:

1. Known allergy to MMAE conjugate of recombinant humanized anti-HER2 monoclonal antibody for injection;
2. Clinical symptoms or diseases of the heart that are not well controlled, such as heart failure of grade 2 or above; b. Unstable angina pectoris; c. Myocardial infarction within 1 year; d. Clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention;
3. There are contraindications for the use of bevacizumab such as severe active bleeding, severe arteriovenous thrombosis events, gastrointestinal obstruction and perforation, and uncontrolled hypertension
4. Major surgical treatment, open biopsy, or significant traumatic injury was received within 28 years prior to treatment
5. In the investigator's judgment, subjects had other factors that might have led to the termination of the study, such as other serious medical conditions (including mental illness) requiring concomitant treatment, serious laboratory abnormalities, and family or social factors that might have affected subjects' safety or the collection of data and samples.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-20 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | From Baseline to disease progress, up to 18 months
  Objective Response Rate was defined as the proportion of patients with a best objective response of complete response (CR) or partial response (PR) according to RECIST criteria (version 1.1)

SECONDARY OUTCOMES:
Progression free survival | From Baseline to primary completion date, about 2 years
  Progression-free survival is defined as the time from enrollment to the first documented disease progression according to RECIST version 1.1, or to death from any cause, whichever occurred first
Overal survival | From Baseline to primary completion date, about 5 years
  Time from randomization to death (from any cause)

CONTACTS AND LOCATIONS:
Overall Officials: Ying Yuan, Study Chair — The Second Affiliated Hospital of Medical College of Zhejiang University
Locations (1):
- The second affiliated hospital of Zhejiang University, Hangzhou, Zhejinag, China